CLINICAL TRIAL: NCT00677157
Title: Evaluation and Diagnosis of Potential Research Subjects With Pain and Fatigue Syndromes
Brief Title: Evaluation and Diagnosis of People With Pain and Fatigue Syndromes
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080132; 08-NR-0132
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Fatigue
Keywords: Fatigue; Fibromyalgia; Pain; Complex Regional Pain Syndrome; Reflex Sympathetic Dystrophy
MeSH Terms: conditions — Fatigue; Fibromyalgia; Pain; Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- screening: participants evaluated for possible inclusion in a natural history or intervention protocol

SUMMARY:
This study will examine people who have pain or fatigue symptoms with a known or unknown diagnosis to determine eligibility for other research studies. No treatment is offered under this protocol.

People 18 years of age or older with symptoms of pain and fatigue may be eligible for this study. Participants undergo standard examinations needed to diagnose or evaluate their symptoms. The results of the test are used to screen subjects for possible participation in other Nursing Institute studies. The study requires from one to three visits at NIH over 12 months for procedures that may include the following:

* Medical history, physical examination and questionnaires related to symptoms and quality of life.
* Blood tests
* Electrocardiogram
* Tender point testing. Pressure is applied to areas of the shoulder, hip, neck, chest, elbow and knee to identify tenderness.

DETAILED DESCRIPTION:
This screening protocol is designed to facilitate patient recruitment to the National Institute of Nursing Research (NINR) clinical research studies on pain and fatigue syndromes. This protocol will also validate the newly developed Saligan Fatigue Questionnaire. Patients must meet the specific requirements of an IRB-approved research study; this protocol serves as a first step for evaluating patients for possible inclusion in a natural history or intervention protocol.

Candidates will be screened with medical history/physical examination, routine laboratory tests, and questionnaires. The physical examination may include the standardized tender point assessment as specified in the American College of Rheumatology (ACR) to diagnose fibromyalgia, measurements of pain (allodynia, hyperalgesia, and hyperpathia), edema, autonomic dysfunction (altered skin color, temperature, or sudomotor activity), and extent of musculoskeletal dysfunction. It will also assess the patients level of pain, fatigue, and quality of life by providing questionnaires for the patients to complete. When the screening is completed, patients will be informed of their options to participate in other NINR interventional or observational clinical research studies. Patients who are not eligible for these studies will be informed of alternative treatments. No treatment is offered under this protocol. Information collected in this protocol will be used to determine eligibility to other NINR protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, patients must meet all of the following:

* Are greater than or equal to 18 years of age;
* Have symptoms of pain and/or fatigue.

EXCLUSION CRITERIA:

Patients with any one of the following will be excluded:

* Inability to provide informed consent for the study;
* Are unwilling or unable to cooperate with the study procedures or travel to NIH for the procedures.

In addition to the above criteria, participants with the following conditions will be excluded from the participating in the peak exercise testing:

* Pregnant or lactating women.
* Unable to refrain from smoking at least 4 hours prior to exercise testing sessions.
* Any medical condition that limits exercise performance and/or affects participants safety during exercise. This includes diseases of the cardiovascular, pulmonary, neurological, metabolic or musculoskeletal systems such as:

  * Diagnosis or history of ischemic heart disease
  * Dilated or hypertrophic cardiomyopathy
  * Non-idiopathic cardiomyopathy
  * Uncontrolled hypertension, defined as a resting blood pressure above 140/90 mmHg
  * Diagnosis or history of right or left-sided heart failure or pulmonary hypertension
  * Diagnosis or history of restrictive or obstructive lung disease
  * Diagnosis or history of stroke
  * Uncontrolled Type I or Type II Diabetes Mellitus
  * Diagnosis of chronic liver disease, chronic kidney disease, acute kidney injury or acute liver failure
  * Metastatic cancer active within the previous five years
  * Mitochondrial disease
  * On medications that would influence aerobic capacity or treadmill performance such as beta-blockers or antiretroviral therapy
  * Active substance abuse including ETOH
  * Medical or psychological instability such that subjects could not reasonably be expected to fulfill the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants for this study will be recruited from a population of patients with pain and fatigue symptoms from other institutes and from referrals from outside centers
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2008-05-23 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Eligibility for participation in NINR study | screening visit
  Qualification for an active NINR study.

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-NR-0132.html